CLINICAL TRIAL: NCT01551303
Title: Effect of Intranasal Neuropeptide on Emotion Perception in Trait Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth A. Hoge, MD, Assistant Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2009P-000387
Record Dates: First submitted 2012-02-21; First posted 2012-03-12 (Estimated); Results first posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-03

CONDITIONS: Social Intelligence
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matched nasal spray placebo.
  Interventions: Drug: Placebo
- Oxytocin (Experimental): Liquid intranasal oxytocin administered in a nasal spray.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Liquid metered-dose nasal spray, 30 IUs, administered once.
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebo — Matched nasal spray placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn more about how emotional processing may be affected by a hormone called oxytocin. Oxytocin is a hormone that occurs naturally in the body, and may play an important role in the way that the brain perceives information.

DETAILED DESCRIPTION:
Extensive research has been conducted to examine cognitive styles in anxiety disorders that may contribute to the psychopathology of these disorders. One of the most consistent findings has been that anxious subjects attend preferentially to threatening stimuli. This attentional bias, which would increase time spent attending to and processing threatening stimuli such as words, sentences, or faces, is thought to help provoke and maintain anxiety states. This is supported by research that demonstrates that reduction in anxiety symptoms is associated with a decrease in attentional bias. Related to an attentional bias is the concept of a perceptual bias, from which people with anxiety disorders may be more perceptive to negative emotional cues. For example, Duncan and Barrett (2007) found a negative correlation between objective awareness of quickly presented faces depicting fear and extraversion. Participants who reported greater extraversion (i.e., pleasure derived from social interactions) were less likely to see 16 ms presentations of faces depicting fear. Thus, it appears that how someone feels is related to and may influence the information they see in their environment. The investigators thus hypothesize that the presence of chronic anxiety disorders may be linked to perceptual biases, and may actually influence how and what information they perceive (their sensory experience). People with anxiety disorders may be less likely to see positive objects and more likely to see negative objects. Although the neurobiological mechanisms underlying these anxiety disorders remain uncertain, one hypothesis implicates the dysregulation of the neuropeptide oxytocin.

Oxytocin is a nine-amino-acid peptide which has a role in maintaining social behavior, and it has been found to decrease anxiety. Researchers have postulated that the anti-anxiety affects of oxytocin are related to the trust and pro-approach behaviors associated with this peptide. For example, mice treated with oxytocin spend more time in the previously avoided open areas of a maze. In a study in humans using healthy volunteers, participants were administered oxytocin or placebo before they played a game with monetary rewards involving trust with a stranger. Those who received oxytocin transferred higher amounts of money to the other player than those who received placebo. This behavior, involving increased comfort with a novel individual or setting, appears to be related to the effects of oxytocin.

As described above, individuals with high levels of anxiety have a perception bias towards emotional stimuli, such as pictures of faces. Oxytocin's anxiolytic, pro-approach and trust effects may decrease this bias, and may cause an individual to experience people or things in the environment as less threatening.

ELIGIBILITY:
Inclusion Criteria:

* No current Axis I according to Diagnostic & Statistical Manual for Psychiatry-IV excluded diagnoses as determined by MINI or Structured Clinical Interview for Diagnosis psychiatric diagnostic interview completed within the past 6 months
* Age 18 to 65
* Subjects must be able to give informed consent and be willing and able to comply with study procedures.

Exclusion Criteria:

* Patients with severe unstable medical illness, clinically significant laboratory findings, or serious medical illness for which hospitalization may be likely within the next three months
* Pregnant or lactating women.
* Subjects currently taking hormones, such as estrogen.
* Known hypersensitivity to oxytocin or to any of the excipients of Syntocinon Nasal spray.
* Known hyponatremia or concurrent use of diuretics.
* Subjects with a history of seizure disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Hoge, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Center for Anxiety and Traumatic Stress Disorders (CATSD), Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults aged 18 to 65 were recruited to the Massachusetts General Hospital through local email and print media advertising from March 2011 to September 2011.
Pre-assignment Details: No enrolled participants were excluded before group assignment.
Groups:
- Oxytocin: Oxytocin, 30 IU in 0.77 ml, intranasal
- Placebo: Placebo, 0.77 ml, intranasal
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started | 25 | 22
Completed | 21 | 15
Not Completed | 4 | 7
Not completed — failed awareness check on vision test | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 25 | 22 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.24 (11.61) | 44.50 (9.62) | 43.30 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 25 | 22 | 47

OUTCOME MEASURES:

1. Primary Outcome: Affective Ratings in Affective Learning Task
Description: We will measure the effect of the drug on affective learning, using the Affective Learning Task. Participants viewed 30 neutral faces, each paired with one sentence describing a negative positive, or neutral behavior, counterbalanced across participants. During the test phase, participants will rate the faces as negative, neutral, or positive. These ratings were averaged. Responses were coded as: negative = -1, neutral = 0, positive =1, so the averaged scores have a possible range between -1 and 1. Since this is not a treatment study for a disease, there is so "better" or "worse" outcome.
Time Frame: 30 minutes after drug administration
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 25 | 22
units on a scale | -0.096 (0.05) | -0.12 (0.054)

ADVERSE EVENTS:
Arm/Group | Placebo | Oxytocin
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 0/22 | 1/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | Oxytocin (N=25)
irritation of nasal passages, temporary (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No